CLINICAL TRIAL: NCT00397241
Title: 24-hour IOP With DTFC and LTFC Monotherapies and the Adjunctive Therapy of DTFC and Latanoprost in Open-angle Glaucoma Insufficiently Controlled With Latanoprost Monotherapy.
Brief Title: 24-hour Study of Dorzolamide/Timolol and Latanoprost/Timolol Fixed Combinations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A733
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — dorzolamide-timolol combination; Latanoprost; Timolol; dorzolamide; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Drug: dorzolamide/timolol
Drug: Drug: latanoprost/timolol
Drug: dorzolamide/timolol and latanoprost
Drug: placebo (artificial tears)

SUMMARY:
The primary objective of this crossover trial is to compare the 3-month mean 24-hour intraocular pressure (IOP) control and safety of dorzolamide/timolol fixed combination (DTFC) given twice daily, versus latanoprost/timolol fixed combination (LTFC) given in the evening and placebo given in the morning, versus adjunctive therapy with DTFC given twice daily and latanoprost 0.005% given once in the evening in open-angle glaucoma patients who are insufficiently controlled with latanoprost monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive primary open-angle (POAG) and exfoliative glaucoma (XFG) patients will be recruited.
* Patients included will be older than 29 years
* Have early to moderate POAG, or XFG (less than 12 mean deviation visual field loss attributed to glaucoma and 0.8 or better vertical cup-to-disc ratio)
* Will be on therapy with latanoprost for more than 3 months;
* Have at treated baseline IOP at 10:00 (two consecutive readings) greater than 21 mm Hg
* Have a reliable visual field (at least two visual fields with less than 30% fixation losses, false positives or negatives)
* Have a best corrected distance Snellen visual acuity > 1/10
* Have corneal pachymetry within the 550 ± 55 μm range, understand the study instructions and are willing to attend all follow-up appointments
* Are willing to comply with study medication usage
* And have open, normal appearing angles

Exclusion Criteria:

* Patients will be excluded if they have: a risk for significant deterioration during the study
* Known previous history of lack of adequate response (< 10% reduction) to any topical glaucoma medication
* Less than 20% daytime IOP reduction on latanoprost;
* Systemic contraindications to topical beta-blockers (asthma, bradycardia, severe congestive heart disease)
* Known contraindications to prostaglandins, history of ocular herpetic disease, or cystoid macular edema
* History of trauma, inflammation, surgery or past use of steroids (within two months)
* Severe dry eyes
* Use of contact lenses
* Signs of ocular infection, except blepharitis
* Corneal abnormality that may affect IOP measurements
* Unwillingness to accept the risk for hyperchromia of the iris or development of hypertrichosis
* And females of childbearing potential or lactating mothers

Ages: 29 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
24-hour IOP control with DTFC will be statistically similar with LTFC given once each evening and placebo in the morning.
Adjunctive therapy with DTFC and latanoprost will provide significantly better 24-hour IOP control than both fixed combinations alone (DTFC and LTFC).

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios GP Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, A University Department of Ophthalmology, AHEPA Hospital, Thessaloniki, Greece
Locations (1):
- Glaucoma Unit, A University Dept of Ophthalmology, Thessaloniki, Greece